CLINICAL TRIAL: NCT04698213
Title: Phase II Study of Avelumab Plus Intermittent Axitinib in Previously Untreated Patients With Metastatic Renal Cell Carcinoma (Tide-A Study)
Brief Title: Avelumab Plus Intermittent Axitinib in Previously Untreated Patients With Metastatic Renal Cell Carcinoma
Acronym: TIDE-A
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIDE-A
Record Dates: First submitted 2019-10-15; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Renal Carcinoma Metastatic
Keywords: metastatic; renal; carcinoma; avelumab; axitinib
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma | interventions — Axitinib; avelumab

STUDY DESIGN:
Intervention Model Description: This is a phase II trial with a partial treatment discontinuation design in patients who achieved tumor decrease greater than 30% compared to baseline during the first 36 weeks of therapy.
  All patients enrolled in the trail will receive axitinib at 5 mg BID plus avelumab at 10 mg/Kg every two weeks.
  Treatment will be continued until progression of disease during the first 36 weeks of therapy. At week 36, patients achieving a tumor decrease ≥ 30% will discontinue axitinib and continue avelumab until progression of disease defined as ≥ 20% increase compared to the tumor burden measured at week 36. At disease progression, axitinib will be restarted at the same dosage used before discontinuation for at least 24 weeks if progression did not occur before. Patients who achieved again tumor decrease of ≥ 30% after 24 weeks of therapy rechallenge with axitinib and avelumab may discontinue axitinib and maintain avelumab until progression of disease in an intermittent manner.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intermittent axitinib plus Avelumab (Experimental): All patients enrolled in the trail will receive axitinib at 5 mg BID plus avelumab at 10 mg/Kg every two weeks.
  Treatment will be continued until progression of disease during the first 36 weeks of therapy. At week 36, patients achieving a tumor decrease ≥ 30% will discontinue axitinib and continue avelumab until progression of disease defined as ≥ 20% increase compared to the tumor burden measured at week 36. At disease progression, axitinib will be restarted at the same dosage used before discontinuation for at least 24 weeks if progression did not occur before. Patients who achieved again tumor decrease of ≥ 30% after 24 weeks of therapy rechallenge with axitinib and avelumab may discontinue axitinib and maintain avelumab until progression of disease in an intermittent manner.
  Interventions: Drug: Axitinib Oral Tablet; Drug: Avelumab

INTERVENTIONS:
Drug: Axitinib Oral Tablet — Axitinib is an orally bioavailable tyrosine kinase inhibitor currently approved in EU for treatment of patients affected by metastatic renal cell carcinoma (mRCC) progressed after another anti VEGFR-tyrosine kinase inhibitor (TKI).
  Axitinib inhibits the proangiogenic cytokines vascular endothelial growth factor (VEGF) and platelet-derived growth factor receptor (PDGF), thereby exerting an anti-angiogenic effect.
Drug: Avelumab — Avelumab is a human immunoglobulin G1 (IgG1) monoclonal antibody directed against the human immunosuppressive ligand programmed death-ligand 1 (PD-L1) protein, with potential immune checkpoint inhibitory and antineoplastic activities. Upon administration, avelumab binds to PD-L1 and prevents the interaction of PD-L1 with its receptor programmed cell death protein 1 (PD-1). This inhibits the activation of PD-1 and its downstream signaling pathways. This may restore immune function through the activation of cytotoxic T lymphocytes (CTLs) targeted to PD-L1-overexpressing tumor cells. In addition, avelumab induces an antibody-dependent cellular cytotoxic (ADCC) response against PD-L1-expressing tumor cells. PD-1, a cell surface receptor belonging to the immunoglobulin superfamily expressed on T cells, negatively regulates T-cell activation and effector function when activated by its ligand, and plays an important role in tumor evasion from host immunity.

SUMMARY:
This study aims to test if patients achieving a tumor response with the combination of axitinib plus avelumab, can discontinued the axitinib in order to delay the resistance to the anti VEGFR-TKI and decrease the related toxicity of the combination therapy.

DETAILED DESCRIPTION:
Axitinib is an orally bioavailable tyrosine kinase inhibitor currently approved in EU for treatment of patients affected by metastatic renal cell carcinoma (mRCC) progressed after another anti VEGFR-tyrosine kinase inhibitor (TKI).

Axitinib inhibits the proangiogenic cytokines vascular endothelial growth factor (VEGF) and platelet-derived growth factor receptor (PDGF), thereby exerting an anti-angiogenic effect.

Avelumab is a human immunoglobulin G1 (IgG1) monoclonal antibody directed against the human immunosuppressive ligand programmed death-ligand 1 (PD-L1) protein, with potential immune checkpoint inhibitory and antineoplastic activities. Upon administration, avelumab binds to PD-L1 and prevents the interaction of PD-L1 with its receptor programmed cell death protein 1 (PD-1). This inhibits the activation of PD-1 and its downstream signaling pathways. This may restore immune function through the activation of cytotoxic T lymphocytes (CTLs) targeted to PD-L1-overexpressing tumor cells. In addition, avelumab induces an antibody-dependent cellular cytotoxic (ADCC) response against PD-L1-expressing tumor cells. PD-1, a cell surface receptor belonging to the immunoglobulin superfamily expressed on T cells, negatively regulates T-cell activation and effector function when activated by its ligand, and plays an important role in tumor evasion from host immunity. PD-L1, a transmembrane protein, is overexpressed on a variety of tumor cell types and is associated with poor prognosis.

The combination of axitinib plus avelumab has been recently reported to be better than sunitinib alone for treatment of previously untreated mRCC patients (Motzer RJ, et al. NEJM 2019). The study reported a median PFS of 13.8 for the combination of axitinib plus avelumab compared to 8.4 months for sunitinib (p<0.001).

To improve the treatment related toxicity, a previous study suggests that the discontinuation of the TKI in patients achieving a tumor response may lead to a longer definitive progression free survival (22.4 months) and overall survival (34.8 months) with a better safety profile (Ornstein MC et al. JCO 2017). Despite the new response to TKI after its reintroduction, the majority of patients progressed after the first months of treatment discontinuation suggesting the necessity to maintain the tumor response.

This study aims to test if patients achieving a tumor response with the combination of axitinib plus avelumab, can discontinued the axitinib in order to delay the resistance to the anti VEGFR-TKI and decrease the related toxicity of the combination therapy.

This is a phase II trial with a partial treatment discontinuation design in patients who achieved tumor decrease greater than 30% compared to baseline during the first 36 weeks of therapy.

All patients enrolled in the trail will receive axitinib at 5 mg BID plus avelumab at 10 mg/Kg every two weeks.

Treatment will be continued until progression of disease during the first 36 weeks of therapy. At week 36, patients achieving a tumor decrease ≥ 30% will discontinue axitinib and continue avelumab until progression of disease defined as ≥ 20% increase compared to the tumor burden measured at week 36. At disease progression, axitinib will be restarted at the same dosage used before discontinuation for at least 24 weeks if progression did not occur before. Patients who achieved again tumor decrease of ≥ 30% after 24 weeks of therapy rechallenge with axitinib and avelumab may discontinue axitinib and maintain avelumab until progression of disease in an intermittent manner.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in this study.

1. Histologically or cytologically confirmed advanced RCC with predominantly clear-cell subtype with primary tumor resected.
2. Male or female subjects aged ≥ 18 years
3. At least one measurable lesion as defined by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
4. Eastern Cooperative Oncology Group performance status 0 or 1.
5. Adequate organ and bone marrow function based upon meeting all of the following laboratory criteria within 10 days before the start of treatment:

   I. Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 GI/L). II. Platelets ≥ 100,000/mm3 (≥ 100 GI/L). III. Hemoglobin ≥ 9 g/dL (≥ 90 g/L). IV. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × upper limit of normal.

   V. Total bilirubin ≤ 1.5 × the upper limit of normal. For subjects with Gilbert's disease ≤ 3 mg/dL (≤ 51.3 µmol/L).

   VI. Serum creatinine ≤ 2.0 × upper limit of normal or calculated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockroft-Gault.
6. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
7. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for at least 30 days after the last dose of study treatment.
8. Negative serum or urine pregnancy test at screening for women of childbearing potential.

Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons. A lactating woman should be advised to not to breastfeed during treatment and for at least one month after the last dose of avelumab.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Prior treatment with systemic therapy for advanced RCC
2. Prior adjuvant or neoadjuvant therapy
3. Bulky or symptomatic disease or hepatic metastases.
4. Prior treatment with any agent specifically targeting T-cell co-stimulation or checkpoint pathways
5. Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis
6. Diagnosis of any non-RCC malignancy occurring within 2 years prior to the date of the start of treatment except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix or low-grade prostate cancer (≤pT2,N0; Gleason 6) with no plans for treatment intervention.
7. Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before the start of treatment. Systemic treatment with radionuclides within 6 weeks before the start of treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
8. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before the start of treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the start of treatment.
9. Concomitant anticoagulation at therapeutic doses with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors).
10. In past 6 months: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack.
11. Chronic treatment with corticosteroids or other immunosuppressive agents (with the exception of inhaled or topical corticosteroids or corticosteroids with a daily dosage equivalent ≤ 10 mg prednisone if given for disorders other than renal cell cancer). Subjects with brain metastases requiring systemic corticosteroid are not eligible.
12. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    I. Cardiovascular disorders:
    1. Symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmias.
    2. Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
    3. Stroke (including TIA), myocardial infarction, or other ischemic event, or thromboembolic event (eg, pulmonary embolism) within 6 months before the start of treatment.

    II. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:
    1. Tumors invading the GI-tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction.
    2. Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before the start of treatment. Note: Complete healing of an intra-abdominal abscess must be confirmed before the start of treatment.

    III. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 3 months before the start of treatment.

    IV. Cavitating pulmonary lesion(s) or known endobronchial disease manifestation.

    V. Lesions invading major pulmonary blood vessels.

    VI. Other clinically significant disorders such as:
    1. Active infection requiring systemic treatment, infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)- related illness, or chronic hepatitis B or C infection (Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening [positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive]).
    2. Serious non-healing wound/ulcer/bone fracture.
    3. Malabsorption syndrome.
    4. Uncompensated/symptomatic hypothyroidism.
    5. Moderate to severe hepatic impairment (Child-Pugh B or C).
    6. Requirement for hemodialysis or peritoneal dialysis.
    7. History of solid organ transplantation including allogenic stem-cell transplantation.
    8. In past 6 months: pulmonary embolism.
13. Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 3 months before the start of treatment. Complete wound healing from major surgery must have occurred 1 month before the start of treatment and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before the start of treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
14. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 msec within 1 month before the start of treatment (see Section 5.5.4 for Fridericia formula). Three ECGs must be performed. If the average of these three consecutive results for QTcF is ≤ 500 msec, the subject meets eligibility in this regard.
15. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
16. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
17. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
18. Has a history of substance abuse or medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
19. Has illness or medical conditions that are unstable or could jeopardize the safety of the patient and his or her compliance in the study.
20. Pregnant or lactating females.
21. Inability to swallow tablets or capsules.
22. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE Grade ≥ 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From the date of the first study drugs administration until week 44
  Evaluate the rate of patients who have a partial response (PR) or complete response (CR) to the study treatment according to RECIST V. 1.1 criteria, as determined by investigator's assessments, at week 8 from axitinib discontinuation and avelumab maintenance, after 36 weeks of induction treatment with the combination of avelumab and axitinib.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years from the last patient first visit (LPFV)
  Will be performed the analyses of Progression free survival in the overall population. PFS, determined using the Kaplan-Meier method, is defined as the time from the first study drugs administration to the date of the first documentation of objective progression of disease (PD) or death due to any cause, whichever occurs first. PFS is calculated according to the RECIST V. 1.1 criteria, as determined by investigator's assessments.
  NB: as per study design, the only PD that causes EoT is the one that occurs during the combined treatment of avelumab and axitinib.
Overall Response Rate (ORR) | 2 years from the last patient first visit (LPFV)
  ORR defined as the rate of patients who have a partial response (PR) or complete response (CR) to the study treatment according to RECIST V. 1.1 criteria as determined by investigator's assessments. The study tumor assessment will be performed every 12 weeks during the combined administration of axitinib and avelumab; during the avelumab maintenance tumor assessment will be performed every 8 weeks for 6 months, then every 12 weeks. NB: as per study design, the only PD that causes EoT is the one that occurs during the combined treatment of avelumab and axitinib.
Disease Control (DC) | 2 years from the last patient first visit (LPFV)
  Disease control (DC) is defined as complete response (CR), partial response (PR), or stable disease (SD) according to the RECIST v.1.1 recorded from enrollment until disease progression assessed by BICR or death due to any cause. DC at 24 weeks is defined as CR, PR or SD ≥24 weeks after enrollment and prior to disease progression assessed by BICR or death due to any cause.
  The DC rate (DCR) and DCR at 24 weeks will be estimated by dividing the number of patients with CR, PR, or SD overall or ≥24 weeks by the number of patients enrol. The corresponding exact 2-sided 95% CIs for DCR and DCR at 24 weeks will be provided.
Overall Survival (OS) | From enrollment date until the date of death due to any cause, assessed up to 5 years
  Overall Survival (OS) is defined as the time from date of enrollment to date of death due to any cause. Patients last known to be alive will be censored at date of last contact. In addition, OS will be tested at the OS final analysis. OS time associated will be summarized using the Kaplan-Meier method and displayed graphically where appropriate. Confidence intervals (CIs) for the 25th, 50th and 75th percentiles will be reported.
Incidence of Treatment-Emergent Adverse Events, Serious adverse events and events of clinical interest, as assessed by the Investigators | From the date of the first study drugs administration up to 90 days after the last dose of study drugs administration
  The primary safety analysis will include all patients who receive at least 1 dose of study drugs and who experienced toxicities as defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 criteria. Safety will be assessed by quantifying the toxicities and grades experienced by subjects who have received the combination avelumab-axitinib and the avelumab alone, including serious adverse events (SAEs) and events of clinical interest (ECIs). Safety will be assessed by reported AEs, SAEs and AESIs according to NCI CTCAE version 5.0. evaluating treatment administration/compliance and safety.
Patient reported outcome (PRO) - Health status | From the enrollment date until the date of first documented progression (that per protocol causes the end of treatment), assessed up to 4 years
  To evaluate the health status of the subjects during the study treatment the "5-Level EuroQol Group's 5-Dimension" (EQ-5D-5L) questionnaire will be administered to the patients within 3 days prior the first study treatment, the first day of each odd cycle (1, 3, 5, etc.) of avelumab, prior to treatment administration, and at the end of treatment visit.
  This questionnaire consists of 2 parts, the EQ-5D index (or simply EQ-5D) and EQ-VAS. The EQ-5D comprises 5 dimensions of health (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression). A unique EQ-5D health state is defined by combining one level from each of the 5 dimensions and is converted to a single summary index or health utility value. The EQ-VAS is a visual analog scale where the patient indicates how good or bad his health is today by marking an appropriate point on a line between 0 to 100, which correspond to the worst and best imaginable health states.
Patient reported outcome (PRO) - Life Status | From the enrollment date until the date of first documented progression (that per protocol causes the end of treatment), assessed up to 4 years
  To evaluate the quality of life of the subjects during the study treatment the "National Comprehensive Cancer Network/ Functional Assessment of Cancer Therapy (FACT)-Kidney Symptom Index 19" (NCCN-FACT FKSI-19) questionnaire will be administered to the patients within 3 days prior the first study treatment, the first day of each odd cycle (1, 3, 5, etc.) of avelumab, prior to treatment administration, and at the end of treatment visit.
  In this questionnaire the score range is 0-76, a score of "0" is a severely symptomatic patient and the highest possible score is an asymptomatic patient.

OTHER OUTCOMES:
Immunohistochemistry expression of markers on tumor tissue | 2 years from the last patient first visit (LPFV)
  Tumor tissue biomarker status at screening phase (ie, positive and negative) will be determined by a predictive biomarker test with an established scoring algorithm defining positive and negative that is developed by the Sponsor; additional tumor tissue biomarkers that may be analyzed include, but may not necessarily be limited to, PD-L1, PBRM1, CD31 expression and quantitation of tumor-infiltrating CD8+ T lymphocytes by IHC.
Expression of a panel of immune-related cytokines and chemokines in blood samples | 2 years from the last patient last visit (LPLV)
  Plasma samples will be collected from enrolled patients at screening phase, after 8 weeks and at End of Treatment. All plasma specimens from each patient will be analysed for the expression of a panel of immune-related cytokines and chemokines. The panel includes interleukin (IL)1b, IL2, IL4, IL5, IL6, IL7, IL8 (CXCL8), IL9, IL10, IL-12p70, IL13, IL15, IL17a, eotaxin, IL1Ra,granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), IFNg, IP10 (CXCL10), monocyte chemoattractant protein (MCP1; CCL2), macrophage inflammatory protein 1a (MIP1a; CCL3), MIP1b (CCL4), TNFa, PDGF-BB, RANTES, tumor necrosis factor a (TNFa), fibroblast growth factor (FGF) and vascular endothelial growth factor (VEGF).
  The plasma markers will be evaluated and analysed considering possible changes. compared to baseline. Each marker (baseline value or at specific timepoint) will be evaluated for a significant correlation to the outcome (i.e. ORR, PFS, OS).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Iacovelli, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (20):
- Italy (20):
  - Azienda Ospedaliera Universitaria di Cagliari- P.O. Duilio Casula Monserrato, Monserrato, Cagliari
  - ASL CN2 Alba-Bra, Alba
  - Irccs Oncologico Istituto Tumori Giovanni Paolo Ii, Bari
  - ASST Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero-Universitaria Di Bologna Suor Orsola Malpighi, Bologna
  - Ospedale Policlinico San Martino, Genova
  - OSPEDALE di LECCE "VITO FAZZI", Lecce
  - Presidio Ospedaliero Unico Av3 - Ospedale Generale Provinciale - Macerata, Macerata
  - Istituto Clinico Humanitas, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Istituti Clinici Scientifici Maugeri, Pavia
  - Irccs Istituto in Tecnologie Avanzate E Modelli Assistenziali in Oncologia Di Reggio Emilia, Reggio Emilia
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
  - Azienda Ospedaliera Santa Maria Terni, Terni
  - Azienda Ospedaliero-Universitaria S. Luigi Gonzaga, Torino
  - Azienda Ospedaliero-Universitaria Integrata Verona - Borgo Roma, Verona

IPD SHARING:
Plan to Share IPD: No